CLINICAL TRIAL: NCT04156035
Title: A Trial to Study Acute and Delayed Effects of a Single Dose of Ketamine on Functional Brain Changes During Emotional/ Cognitive Challenges and at Rest and Their Modulation by Lamotrigine in Healthy Subjects
Brief Title: Ketamine-Induced Brain Changes and Their Modulation by Lamotrigine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Simone Grimm, Prof., Medical School Berlin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MSB-C001
Record Dates: First submitted 2019-10-23; First posted 2019-11-07 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Emotions
MeSH Terms: interventions — Lamotrigine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lamotrigine + Ketamine (Experimental): Pretreatment with lamotrigine will occur 2 hours before the ketamine infusion
  Interventions: Drug: Lamotrigine; Drug: Ketamine
- Placebo + Ketamine (Experimental): Pretreatment with placebo will occur 2 hours before the ketamine infusion
  Interventions: Drug: Ketamine; Drug: Placebo Pretreatment
- Placebo + Placebo (Placebo Comparator): Pretreatment with placebo will occur 2 hours before the placebo infusion
  Interventions: Drug: Placebo Pretreatment; Drug: Placebo Infusion

INTERVENTIONS:
Drug: Lamotrigine — Orally; 300 mg
  Arms: Lamotrigine + Ketamine
Drug: Ketamine — Intravenously; 0.12 mg/kg during the first minute followed by a continuous infusion of approximately 0.31 mg/kg/h over approx. 40 min
  Arms: Lamotrigine + Ketamine; Placebo + Ketamine
Drug: Placebo Pretreatment — Lamotrigine Placebo
  Arms: Placebo + Ketamine; Placebo + Placebo
Drug: Placebo Infusion — Ketamine Placebo
  Arms: Placebo + Placebo

SUMMARY:
This study is firstly designed to investigate acute and delayed effects of a single dose of ketamine on functional brain changes during emotional and cognitive challenges and at rest. Secondly, it aims to investigate whether functional brain changes after ketamine require increased glutamatergic signaling and will accordingly be modulated after pretreatment with lamotrigine.

DETAILED DESCRIPTION:
Despite the rapid antidepressant effects of ketamine, its increasing use as an AD and the recent (2019) FDA approval of ketamine nasal spray as medication for treatment-resistant depression, the exact neurobiological mechanisms underlying its effects remain unclear.

There are numerous reasons, why so far there has been no coherent explanatory framework. Most previous studies focused on investigating a single domain such as functional connectivity (e.g. Deakin et al., 2008; Scheidegger et al., 2012), functional brain changes to either cognitive (e.g. Honey et al., 2005; Driessen et al., 2013) or emotional challenge (e.g. Scheidegger & Grimm et al., 2016; Reed et al., 2019), perfusion (e.g. Pollack et al., 2015), magnetic fields (Salvadore et al., 2010) or neurotransmitter concentrations (e.g. Abdallah et al., 2018). Small sample sizes of as little as 8 subjects, the lack of a control group, the limited number of timepoints for measurement of the above-mentioned parameters, and the failure to modulate glutamatergic signalling after ketamine further limit the informative value of previous findings. What is therefore urgently needed in order to better understand the mechanisms of ketamine, is a study that combines neuroimaging in several modalities, investigates acute as well as delayed effects of ketamine and applies an approach to modulate glutamatergic signaling after ketamine.

Accordingly, this study is designed to investigate acute and delayed effects of a single dose of ketamine on functional brain changes during emotional and cognitive challenge and at rest as well as to investigate the functional significance of increased glutamatergic signalling after ketamine. Measurement of functional brain changes will occur during (acute) and 24 hrs. after a single dose of ketamine, as differential effects are hypothesized. To modulate glutamatergic signaling after ketamine, a lamotrigine pretreatment protocol will be used. It is hypothesized that functional brain changes previously linked to ketamine require increased glutamatergic signaling and will be attenuated by pretreatment with lamotrigine. To test these hypotheses, we will implement a randomized, placebo-controlled, parallel-group design with 3 treatment conditions (lamotrigine + ketamine, placebo + ketamine, placebo + placebo). All subjects will undergo two scanning sessions (acute + post 24 hrs.). In order to include baseline values as covariates in the analyses, imaging will begin 10 minutes before infusion of ketamine/placebo. Pretreatment with lamotrigine or matching placebo will occur 2 hours before the ketamine/placebo infusion. Blood samples will be taken at 0:30, 1:00, 1:30, 2:55 and 4 hours following oral drug administration to determine the plasma pharmacokinetics of lamotrigine, and at 40 minutes after commencing ketamine infusion to confirm target ketamine plasma levels.

ELIGIBILITY:
Main Inclusion Criteria:

* From 18 to 45 years of age, inclusive
* Body Mass Index (BMI) between 18.0 and 28.5 kg/m2, inclusive
* Healthy on the basis of physical examination, medical history, vital signs, clinical laboratory tests, and 12-lead ECG

Main Exclusion Criteria:

* Clinically relevant allergy or drug hypersensitivity
* A history of psychiatric or neurologic disorders
* Alcohol or substance dependence within the last 12 months from screening
* A positive urine drug screen at any visit
* MR exclusion criteria, elevated intracranial pressure or glaucoma
* Hypertonia, cardiac insufficiency, myocardial infarct within last 6 months
* Liver or renal function disorder
* Prescription of psychotropic medication within 28 days prior to screening
* Non-prescription medication, including analgesics and supplements such as vitamins and herbal supplements within 48 hours prior to the baseline visit

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Functional brain changes induced by emotional and cognitive challenge | Measurements will occur during (acute) and 24h after (delayed) a single dose of ketamine
  The primary endpoints of efficacy are the functional brain changes induced by emotional and cognitive challenge during ketamine infusion as compared to placebo and to the responses during ketamine infusion after Lamotrigine pretreatment during and after (post 24 hrs.) in following brain regions (bilateral):
  * Amygdala
  * Hippocampus
  * Dorsolateral Prefrontal Cortex
  * Anterior cingulate Cortex
  * Insula

SECONDARY OUTCOMES:
Changes in resting- state functional connectivity in default- mode network (DMN) and affective network (AN) | Measurements will occur at baseline, during and 24h after a single dose of ketamine
  Changes in resting- state functional connectivity in default- mode network (DMN) and affective network (AN) in the following brain regions (bilateral): Amygdala, Hippocampus, Dorsolateral Prefrontal Cortex, Anterior cingulate Cortex and Insula. During the resting state scan, During this scan, subjects are asked to relax and to keep their eyes open.
Changes in cerebral blood flow in predefined brain regions | Measurements will occur during and 24h after a single dose of ketamine
  Changes in cerebral blood flow (ASL) in in the following brain regions (bilateral): Amygdala, Hippocampus, Dorsolateral Prefrontal Cortex, Anterior cingulate Cortex and Insula. During ASL, subjects engage in no special task, but are asked to close their eyes and relax. ASL provides quantitative parametric images of tissue perfusion.
Association between functional brain changes during emotional and cognitive challenge and ketamine- induced dissociative state | Measurements will occur during and 24h after a single dose of ketamine
  Dissociate state will be investiagted using the Dissoziations-Spannungs-Skala akut (DSS-akut, Stiglmayr et al. 2003).
Association between changes in resting- state functional connectivity and ketamine- induced dissociative state | Measurements will occur during and 24h after a single dose of ketamine
  Dissociate state will be investiagted using the Dissoziations-Spannungs-Skala akut (DSS-akut, Stiglmayr et al. 2003).
Blood concentration of lamotrigine | Measurements will occur at baseline as well as 0.30, 1:00, 1:30, 2:55 and 4h following drug administration
  Blood samples are taken to determine citrate plasma concentration of Lamotrigine to assess plasma levels during fMRI assessments.
Blood concentration of ketamine | Measurements will occur approx. 40 minutes after commencing ketamine infusion
  Blood samples are taken to determine citrate plasma concentration of Ketamine to confirm target exposures (plasma levels) during assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Simone Grimm, PhD, Principal Investigator — Medical School Berlin
Locations (1):
- Medical School Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No